CLINICAL TRIAL: NCT02297490
Title: Evaluation of the Utility of an Environmental Exposure Chamber (EEC) for Assessing Efficacy of Specific Immunotherapy (SIT) in Pivotal Clinical Trials
Brief Title: Evaluation of the Utility of an EEC for Assessing Efficacy of SIT in Pivotal Clinical Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to the interim Analysis results indicating a weaker correlation than anticipated and reported by other study groups.
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Collaborators: Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AL1304AV; AL13BP01 (Other: Inflamax Research INC.)
Record Dates: First submitted 2014-11-12; First posted 2014-11-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinoconjunctivitis; Healthy Volunteers
Keywords: Environmental Exposure Chamber; Specific Immunotherapy; SIT; SCIT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment is identical to the active treatment schedule. The placebo-preparation used is identical to the active solution but without any allergen substance in it.
  Interventions: Drug: Placebo
- Allergovit 6-grasses immunotherapy (Experimental): Immunotherapy will be performed for approx. 5 months. 7 injections will be administered at weekly intervals to reach the maintenance dose. However, dosing must be individualised.
  Interventions: Biological: Allergovit 6-grasses

INTERVENTIONS:
Drug: Placebo — Placebo treatment is identical to the active treatment schedule. The placebo-preparation used is identical to the active solution but without any allergen substance in it.
  Other Names: Comparator
  Arms: Placebo
Biological: Allergovit 6-grasses — Immunotherapy will be performed for approx. 5 months. 7 injections will be administered at weekly intervals to reach the maintenance dose. However, dosing must be individualised.
  Other Names: Specific immunotherapy with an allergoid preparation.
  Arms: Allergovit 6-grasses immunotherapy

SUMMARY:
The study will explore how allergy symptoms experienced during the grass pollen season compare to symptoms experienced in the Environmental Exposure Chamber (EEC).

There are 2 treatments in this study. Both treatments are injected under the skin. Allergovit® Grasses works by helping the body's immune system get used to grass-pollen before the grass pollen season begins which may lead to decreased sensitivity and reduced allergy symptoms during the grass season. Placebo treatment does not contain grass pollen mixture, and is not expected to reduce allergic symptoms overtime.

DETAILED DESCRIPTION:
This is a Phase II trial, with a one year observational/baseline phase followed by a one year double-blind placebo-controlled, randomized, treatment phase. Approx. 137 grass pollen-allergic subjects and 20 non-allergic subjects will be enrolled in the baseline phase of the study. The primary objective of the trial is to investigate the relationship between allergy symptoms experienced by subjects (allergic and non-allergic) upon exposure to grass pollen-allergen in the EEC and the allergy symptoms experienced by subjects during the grass pollen season.

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated seasonal allergic rhinitis/rhinoconjunctivitis with or without allergic asthma
* positive skin prick test
* specific IgE ≥ 0.70 kU/L to mixture of grass pollen allergens
* symptom score of at least 4 per day during the week following the peak-pollen count in the baseline season

Exclusion Criteria:

* undergone previous specific immunotherapy with grass pollen allergens in any formulation less than 5 years prior to the screening date
* currently undergoing any sort of immunotherapy, or has ever undergone specific immunotherapy with unknown allergen
* allergens which are expected to interfere with the grass pollen season
* uncontrolled or partly controlled asthma
* patients with contraindications for SIT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Total Symptom Score (TSS) | 1 year
  Analysis of the relationship between different methods of measurement of efficacy of SIT.
  The AUC of the Total Symptom Score (TSS) as primary endpoint assessed in an EEC after preseasonal treatment
Rhinoconjunctivitis Symptom and Medication Score (RC-SMS) | Grass pollen season from March until July (approx. 11 weeks avarage)
  The AUC of the Rhinoconjunctivitis Symptom and Medication Score (RC-SMS) assessed as primary endpoint during the natural grass pollen season (field-based)
Medication-adjusted Rhinoconjunctivitis Symptom Score (ma-RC-SS) | Grass pollen season from March until July (approx. 11 weeks avarage)
  The AUC of the Medication-adjusted Rhinoconjunctivitis Symptom Score (ma-RC-SS) assessed as primary endpoint during the natural grass pollen season (field-based)

SECONDARY OUTCOMES:
Symptoms (by TSS, RC-SMS, ma-RC-SS) in non-allergic subjects | 1 year
  Evaluation of the relationship of symptoms experienced in EEC and natural grass pollen season. Assessment of symptom specificity provoked by EEC in non-allergic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Patel, Dr., Principal Investigator
Locations (1):
- Inflamax Research INC, Mississauga, Ontario, Canada